CLINICAL TRIAL: NCT00903851
Title: A Prospective, Open-label Trial of Lidoderm® (Lidocaine Patch 5%)in Painful Diabetic and Idiopathic Neuropathy.
Brief Title: Lidoderm® (Lidocaine Patch 5%) in Diabetic and Idiopathic Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sr. Director, Clinical R&D, Endo Pharmaceuticals Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3220-005
Record Dates: First submitted 2009-05-15; First posted 2009-05-19 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Lidoderm

ARMS (1):
- (1) Lidoderm (Experimental): (1)Commercially available Lidoderm® (lidocaine patch 5%), up to four patches applied topically 18 hours on, 6 hours off per day to the area of maximal peripheral neuropathic pain
  Interventions: Drug: Lidoderm

INTERVENTIONS:
Drug: Lidoderm — Patients participated in an 8-week treatment period; patients at one site were to continue treatment for the entire 8 weeks while patients at two sites were to terminate treatment after 3 weeks. Commercially available Lidoderm® (lidocaine patch 5%) was provided to each patient with up to four patches applied topically 18 hours on, 6 hours off per day to the area of maximal peripheral neuropathic pain.
  Other Names: Lidocaine Patch 5%

SUMMARY:
Patients with Type I or II diabetes and painful distal symmetric sensorimotor polyneuropathy with dynamic allodynia of the lower extremities, patients with Type I or II diabetes and pain distal symmetric sensorimotor polyneuropathy with no dynamic allodynia of the lower extremities, or patients with idiopathic distal predominantly sensory neuropathy participated in a Phase IV clinical trial to assess the efficacy of lidocaine patches in treating painful diabetic neuropathy or idiopathic distal sensory neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* At Sites 1, 2, and 3 - Had painful diabetic polyneuropathy of 3 or more months duration
* At Site 1 only - Had clinical signs and symptoms of distal predominantly sensory polyneuropathy of 3 or more months duration. Diagnosis of predominantly sensory polyneuropathy were to be confirmed by either nerve conduction studies (large fiber sensory or sensorimotor axonal neuropathy) or by abnormal epidermal innervations on punch skin biopsy (distal leg/proximal thigh) (Herrmann et al., 1999; Holland et al., 1997)
* Had an average daily pain rating for the baseline week of pain ratings equal to 4 or greater on the 0 to 10 numerical pain rating scale
* Had at least 2 hours of moderate or severe pain intensity due to polyneuropathy daily in the immediately prior 3-month period
* Were using stable analgesic drug therapy for at least 1 week (regimen and dosages) prior to screening visit, with the exception of acetaminophen and lidocaine for patients undergoing a punch skin biopsy

Exclusion Criteria:

* Had prior treatment with topical lidocaine, except for use with the punch skin biopsy procedure
* Were currently under treatment with Class I antiarrhythmic agents (such as tocainide and mexiletine)
* Had any other pain more severe than the painful diabetic or idiopathic neuropathy
* Had open skin lesions in the area where the lidocaine patches were to be applied

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2002-04; Primary Completion 2003-06 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline to Week 3 in average pain intensity as measured from patient diaries using Brief Pain Inventory Question 5. | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)

SECONDARY OUTCOMES:
McGill Pain Questionnaire | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)
Other Pain Questions in BPI | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)
Weekly pain intensity/relief measures | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)
Pain duration using questions that assess duration and frequency of pain | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)
Assessment of allodynia | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)
Neuropathy Pain Scale | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)
Assessment of safety was based on AEs, skin assessment, physical examination, vital signs, clinical laboratory data, and plasma lidocaine levels | Visits - V2 (Day 0), V3 (Day 7), V4 (Day 21), V5 (Day 35), V6/EOs (Day 56)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (4):
- United States (4):
  - Birmingham, Alabama
  - Hueytown, Alabama
  - Jacksonville, Florida
  - Rochester, New York